CLINICAL TRIAL: NCT02443077
Title: A Randomized Double-Blind Phase III Study of Ibrutinib During and Following Autologous Stem Cell Transplantation Versus Placebo in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma of the Activated B-Cell Subtype
Brief Title: Ibrutinib Before and After Stem Cell Transplant in Treating Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NCI-2015-00668; NCI-2015-00668 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BMT CTN 1201; A051301; A051301 (Other: Alliance for Clinical Trials in Oncology); A051301 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2025-09-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma Activated B-Cell Type; Refractory Diffuse Large B-Cell Lymphoma Activated B-Cell Type
MeSH Terms: interventions — Bone Marrow Transplantation; Stem Cell Transplantation; Carmustine; Cyclophosphamide; Cytarabine; Etoposide; ibrutinib; Melphalan; Pharmacogenomic Testing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (ibrutinib, chemotherapy, autoHCT) (Experimental): CONDITIONING REGIMEN: Investigators may choose to use either the BEAMi or CBVi regimen.
  BEAMi: Patients receive ibrutinib PO on days -6 to -1 or days -7 to -2 if a day of rest is planned, carmustine IV over 2 hours on day -6, etoposide IV BID over 1-2 hours and cytarabine IV BID over 1-2 hours on days -5 to -2, and melphalan IV over 20-30 minutes on day -1.
  CBVi: Patients receive ibrutinib PO on days -6 to -1 or days -7 to -2 if a day of rest is planned, carmustine IV over 2 hours on day -6, etoposide IV over 4 hours on day -4, and cyclophosphamide IV on day -2.
  TRANSPLANT: In both arms, patients undergo autologous hematopoietic progenitor cell or bone marrow transplant on day 0.
  CONTINUATION REGIMEN: Beginning 30-60 days after transplant, patients receive ibrutinib PO on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Bone Marrow Transplantation; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Etoposide; Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Other: Pharmacogenomic Study
- Arm II (placebo, chemotherapy, autoHCT) (Placebo Comparator): CONDITIONING REGIMEN: Patients receive placebo PO on days -6 to -1 and receive 1 of the 2 conditioning regimens as in Arm I.
  TRANSPLANT: Patients undergo autologous hematopoietic progenitor cell or bone marrow transplant on day 0.
  CONTINUATION REGIMEN: Beginning 30-60 days after transplant, patients receive placebo PO on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression may crossover Arm I.
  Interventions: Procedure: Autologous Bone Marrow Transplantation; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Other: Pharmacogenomic Study; Other: Placebo Administration

INTERVENTIONS:
Procedure: Autologous Bone Marrow Transplantation — Undergo autologous hematopoietic progenitor cells or bone marrow transplant
  Other Names: ABMT; Autologous Blood and Marrow Transplantation; Autologous Bone Marrow Transplant; Autologous Marrow Transplantation
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous hematopoietic progenitor cells or bone marrow transplant
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; NSC 409962; NSC409962; SK 27702; SRI 1720; WR 139021; WR-139021; WR139021
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
  Arms: Arm I (ibrutinib, chemotherapy, autoHCT)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo, chemotherapy, autoHCT)

SUMMARY:
This randomized phase III trial studies ibrutinib to see how well it works compared to placebo when given before and after stem cell transplant in treating patients with diffuse large B-cell lymphoma that has returned after a period of improvement (relapsed) or does not respond to treatment (refractory). Before transplant, stem cells are taken from patients and stored. Patients then receive high doses of chemotherapy to kill cancer cells and make room for healthy cells. After treatment, the stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. Ibrutinib is a drug that may stop the growth of cancer cells by blocking a protein that is needed for cell growth. It is not yet known whether adding ibrutinib to chemotherapy before and after stem cell transplant may help the transplant work better in patients with relapsed or refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the ability of ibrutinib to improve 24-month progression free survival (PFS) compared to placebo in patients with non-germinal center B-cell-like (GCB) diffuse large B-cell lymphoma (DLBCL) as determined by immunohistochemistry (IHC).

SECONDARY OBJECTIVES:

I. To evaluate the ability of ibrutinib to improve overall survival (OS) compared to placebo.

II. To evaluate the ability of ibrutinib to improve progression free survival (PFS) compared to placebo.

III. To evaluate the ability of ibrutinib to improve post-transplant response rates compared to placebo.

IV. To evaluate time to hematopoietic recovery in the two arms. V. To evaluate the safety and tolerability of ibrutinib compared to placebo. VI. To evaluate the incidence of secondary malignancies in the two arms. VII. To evaluate immune reconstitution in the two arms.

CORRELATIVE SCIENCE OBJECTIVES:

I. To assess whether pre-autologous hematopoietic stem cell transplantation (AutoHCT) positive fludeoxyglucose F-18 (FDG)-positron emission tomography (PET) is associated with inferior 24-month PFS as well as PFS and OS.

II. To assess whether pre-AutoHCT FDG-PET results are differentially associated with 24-month PFS, PFS and OS in the ibrutinib versus placebo arms.

III. To evaluate the application of the Lugano criteria and change in quantitative measurements between pre-AutoHCT and post AutoHCT (e.g. delta standard uptake variable [SUV], %SUV decline and %metabolic tumor volume [MTV] decline, and other available applicable quantitative measurements) to assess the association between changes in these variables and outcomes, such as PFS and OS.

IV. To assess whether the GSTT1 null polymorphism is correlated with pulmonary toxicity after BCNU (carmustine)-containing conditioning regimens as part of autologous stem cell transplantation.

V. To assess whether other polymorphisms in the BCNU metabolism pathway or BCNU damage repair pathway(s) are associated with pulmonary toxicity after BCNU-containing conditioning regimens as part of autologous stem cell transplantation.

VI. To evaluate whether any of the proposed deoxyribonucleic acid (DNA) polymorphisms are associated with other toxicities.

VII. To assess whether DLBCL subtype based on the lymphoma subtyping test (LST) is associated with 24-month PFS, PFS, and OS with ibrutinib compared to placebo in patients treated on this protocol.

VIII. To assess whether activating mutations in the BCR pathway are associated with response to ibrutinib and with clinical outcomes in patients treated on this protocol.

IX. To assess whether there are any phenotypic associations with IHC markers (particularly MYC protein expression level) and presence of these mutations.

X. To assess whether BCL2, MYC, and Ki67 expression by IHC affect clinical outcomes in patients treated on this protocol.

XI. To assess whether translocations in MYC with or without BCL2 and BC6 have poor outcomes in patients treated on this protocol and whether ibrutinib modifies the prognosis.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

CONDITIONING REGIMEN:

ARM I: Investigators may choose to use either the BEAMi (carmustine, etoposide, cytarabine, melphalan, ibrutinib) or CBVi (cyclophosphamide, carmustine, etoposide, ibrutinib) regimen.

BEAMi: Patients receive ibrutinib orally (PO) on days -6 to -1, carmustine intravenously (IV) over 2 hours on day -6, etoposide IV twice daily (BID) over 1-2 hours and cytarabine IV BID over 1-2 hours on days -5 to -2, and melphalan IV over 20-30 minutes on day -1. Optionally, if a day of rest is planned, patients may receive BEAMi on days -7 to -2.

CBVi: Patients receive ibrutinib PO on days -6 to -1, carmustine IV over 2 hours on day -6, etoposide IV over 4 hours on day -4, and cyclophosphamide IV on day -2. Optionally, if a day of rest is planned, patients may receive CBVi on days -7 to -2.

ARM II: Patients receive placebo PO on days -6 to -1 and receive 1 of the 2 conditioning regimens as in Arm I.

TRANSPLANT: In both arms, patients undergo autologous hematopoietic progenitor cell or bone marrow transplant on day 0.

CONTINUATION REGIMEN:

ARM I: Beginning 30-60 days after transplant, patients receive ibrutinib PO on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Beginning 30-60 days after transplant, patients receive placebo PO on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression may crossover Arm I.

After completion of treatment, patients are followed up every 6 months for up to 60 months from registration.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION ELIGIBILITY CRITERIA (STEP 0)
* Patients must have paraffin tissue from the diagnostic or relapse biopsy available to be submitted for central pathology review; this review is mandatory prior to registration to confirm eligibility and should be initiated as soon as possible
* ELIGIBILITY CRITERIA (STEP 1)
* Diagnosis of World Health Organization (WHO) diffuse large B-cell lymphoma, non-GCB by central review confirmation
* Patient must be deemed eligible to proceed with high-dose chemotherapy and autologous stem cell transplantation by local transplant center
* New York Heart Association class I or less; ordinary physical activity does not cause undue fatigue, palpitations, dyspnea, or angina pain; patients 60 years or older must have a left ventricular ejection fraction (LVEF) at rest >= 40% measured by echocardiogram or multi-gated acquisition (MUGA)
* Diffusion capacity of the lung for carbon monoxide (DLCO) >= 40% of predicted (corrected or uncorrected for hemoglobin per institutional standards)
* Forced expiratory volume in 1 second (FEV1) >= 40% of predicted (corrected or uncorrected for hemoglobin per institutional standards)
* Forced vital capacity (FVC) >= 40% of predicted (corrected or uncorrected for hemoglobin per institutional standards)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless isolated hyperbilirubinemia attributed to Gilbert's syndrome
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x upper limit of normal (ULN)
* Creatinine =< 2.0 mg/dL OR creatinine clearance (calculated clearance permitted) >= 40 mL/min by Cockcroft-Gault formula
* Prothrombin time (PT)/ international normalized ration (INR) < 1.5 x ULN and partial thromboplastin time (PTT) (activated [a]PTT) < 1.5 x ULN
* Patient must have progressed or be refractory to prior anthracycline-containing chemotherapy (e.g. rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone [R-CHOP], dose adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab [DA-EPOCH-R], etc)
* No more than 3 prior regimens for large cell component (e.g. one induction and two salvage therapies); monoclonal antibody alone or involved field/involved site radiotherapy do not count as lines of therapy. Prior CART therapy is allowed and counts as one line of therapy
* Prior use of ibrutinib is allowed unless patient has had disease progression while receiving ibrutinib
* Patient must have chemosensitive disease as defined by at least a partial response to salvage therapy at their latest assessment
* No major surgery =< 7 days prior to registration and no minor surgery =< 3 days prior to registration (with the exception of intravenous access placement, e.g. Hickman or peripherally inserted central catheter [PICC])
* Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects; therefore, for women of childbearing potential only, a negative serum pregnancy test must be obtained within 14 days prior to registration

  * Women of childbearing potential must use adequate contraception from study start to one month after the last dose of protocol therapy; adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence; men must practice complete abstinence or agree to use an adequate contraception method from study start to one month after the last dose of protocol therapy
* Age >= 18 years
* Patients should not require chronic use of strong CYP3A inhibitors or strong CYP3A inducers
* Patients should not require concurrent therapeutic doses of steroids (> 20 mg of prednisone/day or equivalent) unless they need them for the indications; steroids should be discontinued for 14 days before starting protocol treatment
* Human immunodeficiency virus (HIV) infected patients are eligible provided they meet all other eligibility criteria, and:

  * There is no prior history of acquired immunodeficiency syndrome (AIDS) defining conditions other than historically low CD4+ T-cell count or B-cell lymphoma
  * In the opinion of an expert in HIV disease, prospects for long-term survival are excellent were it not for the diagnosis of lymphoma
  * Use of HIV protease inhibitors as part of the anti-HIV regimen OR as a pharmacologic booster is not allowed
  * Zidovudine is not allowed
  * Once daily combination pills for HIV containing a pharmacologic booster such as cobicistat are not allowed
  * Patients with multi-drug resistant HIV are not eligible
* Patients cannot have:

  * Active central nervous system or meningeal involvement by lymphoma; patients with a history of central nervous system (CNS) or meningeal involvement must be in a documented remission by cerebrospinal fluid (CSF) evaluation and contrast-enhanced magnetic resonance imaging (MRI) imaging for at least 91 days prior to registration
  * Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy
  * A known bleeding diathesis
  * Requirement for warfarin or similar vitamin K antagonists; these drugs are prohibited 28 days prior to the first treatment and throughout the trial
  * History of stroke or intracranial hemorrhage =< 6 months before treatment
  * Currently active, clinically significant hepatic impairment (Child-Pugh class B or C according to the Child Pugh classification
  * History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib or other agents used in study
  * Serologic status reflecting active hepatitis B or C infection; patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment; (PCR positive patients will be excluded)
* Eastern Cooperative Oncology Group (ECOG) performance status must be =< 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2025-12-24 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Charalambos B Andreadis, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (281):
- United States (280):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Ibrutinib, Chemotherapy, autoHCT): CONDITIONING REGIMEN: Investigators may choose to use either the BEAMi or CBVi regimen.> BEAMi: Patients receive ibrutinib PO on days -6 to -1 or days -7 to -2 if a day of rest is planned, carmustine IV over 2 hours on day -6, etoposide IV BID over 1-2 hours and cytarabine IV BID over 1-2 hours on days -5 to -2, and melphalan IV over 20-30 minutes on day -1. > CBVi: Patients receive ibrutinib PO on days -6 to -1 or days -7 to -2 if a day of rest is planned, carmustine IV over 2 hours on day -6, etoposide IV over 4 hours on day -4, and cyclophosphamide IV on day -2.> TRANSPLANT: In both arms, patients undergo autologous hematopoietic progenitor cell or bone marrow transplant on day 0.> CONTINUATION REGIMEN: Beginning 30-60 days after transplant, patients receive ibrutinib PO on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.> Autologous Bone Marrow Transplantation: Undergo autologous hematopoietic progenitor cells or bone marrow transplant> Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous hematopoietic progenitor cells or bone marrow transplant> Carmustine: Given IV> Cyclophosphamide: Given IV> Cytarabine: Given IV> Etoposide: Given IV> Ibrutinib: Given PO> Laboratory Biomarker Analysis: Correlative studies> Melphalan: Given IV> Pharmacogenomic Study: Correlative studies
- Arm II (Placebo, Chemotherapy, autoHCT): CONDITIONING REGIMEN: Patients receive placebo PO on days -6 to -1 and receive 1 of the 2 conditioning regimens as in Arm I.> >>
  TRANSPLANT: Patients undergo autologous hematopoietic progenitor cell or bone marrow transplant on day 0.> >> >> >> > >> >> >> CONTINUATION REGIMEN: Beginning 30-60 days after transplant, patients receive placebo PO on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression may crossover Arm I.> >> >> >> > >> >> >> Autologous Bone Marrow Transplantation: Undergo autologous hematopoietic progenitor cells or bone marrow transplant> >> >> >> > >> >> >> Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous hematopoietic progenitor cells or bone marrow transplant> >> >> >> > >> >> >> Carmustine: Given IV> >> >> >> > >> >> >> Cyclophosphamide: Given IV> >> >> >> > >> >> >> Cytarabine: Given IV> >> >> >> > >> >> >> Etoposide: Given IV> >> >> >> > >> >> >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >>
  >>
  >
  >>
  >>
  >> Melphalan: Given IV>
  >>
  >>
  >>
  >
  >>
  >>
  >> Pharmacogenomic Study: Correlative studies>
  >>
  >>
  >>
  >
  >>
  >>
  >> Placebo Administration: Given PO
- Safety Cohort: AutoHCT + Ibrutinib (Cycle 1)> >> Ibrutinib 560 mg† days -6 to -1>
  >> Ibrutinib Continuation>
  >> (Cycles 2-13)**>
  >> Ibrutinib 560 mg daily
Period: Overall Study
Arm/Group | Arm I (Ibrutinib, Chemotherapy, autoHCT) | Arm II (Placebo, Chemotherapy, autoHCT) | Safety Cohort
Started | 45 | 43 | 6
Crossover | 2 | 0 | 0
Completed | 10 | 9 | 6
Not Completed | 35 | 34 | 0

BASELINE CHARACTERISTICS:
Population: Only randomized arms were analyzed. Safety cohort was excluded per protocol: These patients will not be randomized and will be excluded in the statistical analysis to compare the two arms.
Groups:
- Safety Cohort: AutoHCT + Ibrutinib (Cycle 1) Ibrutinib 560 mg† days -6 to -1 Ibrutinib Continuation (Cycles 2-13)** Ibrutinib 560 mg daily
- Total: Total of all reporting groups
Arm/Group | Arm I (Ibrutinib, Chemotherapy, autoHCT) | Arm II (Placebo, Chemotherapy, autoHCT) | Safety Cohort | Total
Number analyzed (Participants) | 45 | 43 | 6 | 94
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [55 to 67] | 59 [51 to 66] | 52.5 [46 to 64] | 61 [51 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 1 | 41
  Male | 25 | 23 | 5 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 0 | 5
  Not Hispanic or Latino | 43 | 40 | 6 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 4
  White | 38 | 39 | 3 | 80
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 3 | 9
Prior Ibrutinib [Count of Participants; unit: Participants] | 1 | 0 | 0 | 1
Time to relapse [Count of Participants; unit: Participants]
  <= 12 months (includes refractory) | 21 | 21 | 5 | 47
  > 12 months | 24 | 22 | 1 | 47
Type of transplant regimen planned [Count of Participants; unit: Participants]
  BEAM | 42 | 41 | 5 | 88
  CBV | 3 | 2 | 1 | 6
Number of prior lines of chemo [Median (Full Range); unit: chemo lines] | 2 [1 to 3] | 2 [1 to 3] | 2 [2 to 3] | 2 [1 to 3]
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction. > ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. > ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours. > ECOG = 0 is better. ECOG = 2 is worse.
  Participants
    0 | 14 | 18 | 2 | 34
    1 | 27 | 23 | 4 | 54
    2 | 4 | 2 | 0 | 6
LDH [Median (Inter-Quartile Range); unit: U/L] | 251 [178 to 350] | 229.5 [167 to 535] | 292.5 [219 to 366] | 235 [171 to 419]
Refractory Disease [Count of Participants; unit: Participants] | 10 | 8 | 2 | 20
Stage of Disease at Relapse [Count of Participants; unit: Participants] — Stage 1 - Cancer is found in one lymph node, a lymphoid organ such as the thymus or one area of a single organ outside of the lymphatic system.>> Stage 2 - Cancer is found in two lymph nodes (both on the same side of the diaphragm) or extends from one lymph node into a nearby organ.>> Stage 3 - Cancer is found in several lymph nodes, both above and below the diaphragm, and may also have spread to the spleen.>> Stage 4 - Cancer is found outside of the lymphatic system or in two or more distant organs such as the liver or the lungs.>> Stage 1 is better. Stage 4 is worse
  Participants
    I | 3 | 4 | 0 | 7
    II | 11 | 7 | 1 | 19
    III | 11 | 11 | 2 | 24
    IV | 20 | 21 | 3 | 44
Baseline Deauville Score [Count of Participants; unit: Participants] — Deauville 5PS: 1, no uptake above background; 2, uptake ≤ mediastinum; 3, uptake > mediastinum but ≤ liver; 4, uptake moderately > liver; 5, uptake markedly higher than liver and/or new lesions; X, new areas of uptake unlikely to be related to lymphoma.
  Participants
    Score 1-2 | 18 | 12 | 0 | 30
    Score 3-4 | 12 | 11 | 0 | 23
    Score 5 | 3 | 5 | 0 | 8
Extranodal Involvement [Count of Participants; unit: Participants]
  Bone marrow | 7 | 3 | 0 | 10
  Liver | 0 | 1 | 0 | 1
  Lung | 6 | 2 | 0 | 8
  Subcutaneous Tissue | 4 | 1 | 1 | 6
  Pleura | 2 | 0 | 0 | 2
  Spleen | 3 | 3 | 2 | 8
  Other | 9 | 6 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: 24-month Progression-free Survival (PFS), Defined as the Proportion of Patients Who Are Alive and Progression-free 2 Years From Randomization
Description: Will be assessed using the Lugano classification.
Time Frame: Time between registration and disease progression or death, whichever comes first, assessed at 24 months
Population: Participants that completed at least one cycle of treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Arm I (Ibrutinib, Chemotherapy, autoHCT): CONDITIONING REGIMEN: Investigators may choose to use either the BEAMi or CBVi regimen.> BEAMi: Patients receive ibrutinib PO on days -6 to -1 or days -7 to -2 if a day of rest is planned, carmustine IV over 2 hours on day -6, etoposide IV BID over 1-2 hours and cytarabine IV BID over 1-2 hours on days -5 to -2, and melphalan IV over 20-30 minutes on day -1.> CBVi: Patients receive ibrutinib PO on days -6 to -1 or days -7 to -2 if a day of rest is planned, carmustine IV over 2 hours on day -6, etoposide IV over 4 hours on day -4, and cyclophosphamide IV on day -2.> TRANSPLANT: In both arms, patients undergo autologous hematopoietic progenitor cell or bone marrow transplant on day 0.> CONTINUATION REGIMEN: Beginning 30-60 days after transplant, patients receive ibrutinib PO on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.> Autologous Bone Marrow Transplantation: Undergo autologous hematopoietic progenitor cells or bone marrow transplant Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous hematopoietic progenitor cells or bone marrow transplant Carmustine: Given IV Cyclophosphamide: Given IV Cytarabine: Given IV Etoposide: Given IV Ibrutinib: Given PO Laboratory Biomarker Analysis: Correlative studies Melphalan: Given IV Pharmacogenomic Study: Correlative studies
Arm/Group | Arm I (Ibrutinib, Chemotherapy, autoHCT) | Arm II (Placebo, Chemotherapy, autoHCT)
Number analyzed (Participants) | 39 | 38
proportion of participants | 0.576 [0.421 to 0.788] | 0.408 [0.265 to 0.628]

2. Secondary Outcome: Overall Survival (OS)
Description: For each arm, the distribution of OS will be estimated using the Kaplan-Meier method. OS will be compared between the two arms using the log-rank test and Cox regression method adjusting for the known predictors.
Time Frame: The time between randomization and death from any cause, assessed up to 5 years (60 months)
Reporting Status: Not Posted

3. Secondary Outcome: Time to Hematopoietic Engraftment
Description: Will be defined as platelet count greater than or equal to 20,000/uL following nadir.
Time Frame: First day of one week without platelet transfusion, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm I (Ibrutinib, Chemotherapy, autoHCT) | Arm II (Placebo, Chemotherapy, autoHCT)
Number analyzed (Participants) | 39 | 38
days | 14.0 [12.0 to 17.0] | 14.5 [13.0 to 19.0]

4. Secondary Outcome: PFS
Description: For each arm, the distribution of PFS will be estimated using the Kaplan-Meier method. PFS will be compared between the two arms using the log-rank test and Cox regression method adjusting for the known predictors.
Time Frame: Time between registration and disease progression or death, whichever comes first, assessed up to 5 years (60 months)
Reporting Status: Not Posted

5. Secondary Outcome: Response Rate Using the Lugano Classification
Description: The metabolic response proportion following AutoHCT will be compared between the two arms using chi-squared test.
Time Frame: Up to 60 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Ibrutinib, Chemotherapy, autoHCT) | Arm II (Placebo, Chemotherapy, autoHCT)
Number analyzed (Participants) | 39 | 38
proportion of participants | 0.590 [0.421 to 0.744] | 0.553 [0.383 to 0.714]

6. Secondary Outcome: Treatment-related Mortality
Description: Treatment-related mortality will be summarized using contingency tables.
Time Frame: Up to 60 months
Measure: Number; unit: participants
Arm/Group | Arm I (Ibrutinib, Chemotherapy, autoHCT) | Arm II (Placebo, Chemotherapy, autoHCT)
Number analyzed (Participants) | 13 | 12
participants
  Disease-related | 6 | 8
  Infection | 4 | 0
  New Primary | 1 | 0
  Other/Unknown | 2 | 4

7. Secondary Outcome: Incidence of Hematologic Toxicity of Ibrutinib Therapy
Description: Hematologic toxicity will be summarized using contingency tables.
Time Frame: Up to 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Ibrutinib, Chemotherapy, autoHCT) | Arm II (Placebo, Chemotherapy, autoHCT)
Number analyzed (Participants) | 39 | 38
Participants
  Grade 3 Event | 6 | 9
  Grade 4 Event | 13 | 11
  Grade 5 Event | 0 | 0

8. Secondary Outcome: Incidence of Secondary Malignancies
Description: Incidence of secondary malignancies will be summarized using contingency tables.
Time Frame: Up to 60 months
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Ibrutinib, Chemotherapy, autoHCT): CONDITIONING REGIMEN: Investigators may choose to use either the BEAMi or CBVi regimen.>>> >>> BEAMi: Patients receive ibrutinib PO on days -6 to -1 or days -7 to -2 if a day of rest is planned, carmustine IV over 2 hours on day -6, etoposide IV BID over 1-2 hours and cytarabine IV BID over 1-2 hours on days -5 to -2, and melphalan IV over 20-30 minutes on day -1. >>>
  >>> CBVi: Patients receive ibrutinib PO on days -6 to -1 or days -7 to -2 if a day of rest is planned, carmustine IV over 2 hours on day -6, etoposide IV over 4 hours on day -4, and cyclophosphamide IV on day -2.>>>
  >>> TRANSPLANT: In both arms, patients undergo autologous hematopoietic progenitor cell or bone marrow transplant on day 0.>>>
  >>> CONTINUATION REGIMEN: Beginning 30-60 days after transplant, patients receive ibrutinib PO on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.>>>
  >>> Autologous Bone Marrow Transplantation: Undergo autologous hematopoietic progenitor cells or bone marrow transplant>>>
  >>> Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous hematopoietic progenitor cells or bone marrow transplant>>>
  >>> Carmustine: Given IV>>>
  >>> Cyclophosphamide: Given IV>>>
  >>> Cytarabine: Given IV>>>
  >>> Etoposide: Given IV>>>
  >>> Ibrutinib: Given PO>>>
  >>> Laboratory Biomarker Analysis: Correlative studies>>>
  >>> Melphalan: Given IV>>>
  >>> Pharmacogenomic Study: Correlative studies
- Arm II (Placebo, Chemotherapy, autoHCT): CONDITIONING REGIMEN: Patients receive placebo PO on days -6 to -1 and receive 1 of the 2 conditioning regimens as in Arm I.>>> >>> TRANSPLANT: Patients undergo autologous hematopoietic progenitor cell or bone marrow transplant on day 0.>>>
  >>> CONTINUATION REGIMEN: Beginning 30-60 days after transplant, patients receive placebo PO on days 1-28. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression may crossover Arm I.>>>
  >>> Autologous Bone Marrow Transplantation: Undergo autologous hematopoietic progenitor cells or bone marrow transplant>>>
  >>> Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous hematopoietic progenitor cells or bone marrow transplant>>>
  >>> Carmustine: Given IV>>>
  >>> Cyclophosphamide: Given IV>>>
  >>> Cytarabine: Given IV>>>
  >>> Etoposide: Given IV>>>
  >>> Laboratory Biomarker Analysis: Correlative studies>>>
  >>> Melphalan: Given IV>>>
  >>> Pharmacogenomic Study: Correlative studies>>>
  >>> Placebo Administration: Given PO
Arm/Group | Arm I (Ibrutinib, Chemotherapy, autoHCT) | Arm II (Placebo, Chemotherapy, autoHCT)
Number analyzed (Participants) | 39 | 38
Participants | 1 | 0

9. Other Pre Specified Outcome: Fludeoxyglucose Positron Emission Tomography (FDG-PET) Imaging Results
Description: PFS and OS will be compared between PET/computed tomography (CT) positive and negative groups using the two-sample log-rank test with a 2-sided alpha of 5%. A Cox regression model will be conducted to regress PFS and OS on PET/CT positivity. Deauville criteria analyses will be conducted with cutoffs at scores of 2 and 3, and quantitative measurements, e.g. delta standard uptake value (SUV), %SUV decline and %MTV decline, in place of the dichotomous FDG-PET/CT outcome. Positive/negative predictive values, sensitivity and specificity of PET/CT further estimated by dichotomizing the PFS and OS at 2 years.
Time Frame: Baseline
Reporting Status: Not Posted

10. Other Pre Specified Outcome: GSTT1 Null Allele Expression
Description: GSTT1 null allele expression will be associated with carmustine toxicity. Quantified using the standard Common Terminology Criteria for Adverse Events and changes in diffusing capacity of the lungs for carbon monoxide from baseline.
Time Frame: Baseline
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Single-nuclear Polymorphisms (SNPs) in the BCNU Metabolism or Damage Repair Pathways
Description: All SNPs will be evaluated for deviation from Hardy-Weinberg. In the absence of a hypothesized effect, analyses will be powered for allele dosing (i.e., additive) effects. The Cochran-Armitage test (for binary endpoints), Jonkheere-Terpstra test (for quantitative traits including biomarker or gene expressions in serum or tumor ribonucleic acid) and the Cox score test (for censored time-to-event outcomes) will be used to quantify marginal associations. Multivariable models, with molecular, clinical and demographic variables, will be constructed using conditional inference trees and random forests.
Time Frame: Baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: BCR Pathway Mutations
Description: The mutation of CD79a/b, caspase recruitment domain family, member 11 (CARD11), tumor necrosis factor, alpha-induced protein 3 TNFAIP3), and myeloid differentiation primary response 88 (MYD88) will be associated with each outcome in the ibrutinib arm (Arm A) using the chi-squared test for response rate and the log-rank test for each censored outcome. Similar analyses will be conducted for the placebo arm (Arm B) to show that the association between mutation and the outcomes observed in the ibrutinib arm is not observed in the placebo arm.
Time Frame: Baseline
Reporting Status: Not Posted

13. Other Pre Specified Outcome: BCL2, MYC, and Ki67 Expression in Tissue Samples by Immunohistochemistry (IHC)
Description: The expression of BCL2, MYC, and Ki67 will be analyzed to assess whether they affect clinical outcomes.
Time Frame: Baseline
Reporting Status: Not Posted

14. Other Pre Specified Outcome: MYC Translocations
Description: Translocations in MYC with or without BCL2, and BCL6 will be analyzed to determine whether they are related to poor outcomes and whether ibrutinib modifies the prognosis.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 60 months
Groups:
- Crossover Arm: Pharmacogenomic Study: Correlative studies
Arm/Group | Arm I (Ibrutinib, Chemotherapy, autoHCT) | Arm II (Placebo, Chemotherapy, autoHCT) | Safety Cohort | Crossover Arm
All-Cause Mortality (participants affected / at risk) | 14/45 | 10/43 | 3/6 | 2/2
Serious Adverse Events (participants affected / at risk) | 22/45 | 23/43 | 4/6 | 1/2
Other Adverse Events (participants affected / at risk) | 36/45 | 38/43 | 6/6 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Ibrutinib, Chemotherapy, autoHCT) (N=45) | Arm II (Placebo, Chemotherapy, autoHCT) (N=43) | Safety Cohort (N=6) | Crossover Arm (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (7) | 4 (4) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 1 (2) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Ibrutinib, Chemotherapy, autoHCT) (N=45) | Arm II (Placebo, Chemotherapy, autoHCT) (N=43) | Safety Cohort (N=6) | Crossover Arm (N=2)
Anemia (Blood and lymphatic system disorders) | 18 (50) | 9 (20) | 1 (6) | 0 (0)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 5 (11) | 2 (10) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6) | 5 (5) | 2 (2) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (7) | 3 (5) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 5 (10) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (5) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 12 (17) | 12 (21) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 29 (60) | 28 (52) | 6 (8) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 6 (8) | 2 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 27 (59) | 26 (40) | 5 (8) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (18) | 14 (19) | 3 (4) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 4 (11) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 34 (111) | 30 (78) | 6 (13) | 1 (1)
Fever (General disorders) | 18 (21) | 20 (25) | 5 (6) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 2 (8) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 2 (3) | 0 (0) | 1 (3) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 5 (9) | 2 (2) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 6 (13) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (11) | 2 (4) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (10) | 2 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (10) | 2 (2) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 4 (15) | 2 (5) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (13) | 6 (16) | 1 (1) | 1 (2)
Lymphocyte count increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 16 (33) | 15 (21) | 2 (7) | 0 (0)
Platelet count decreased (Investigations) | 18 (46) | 10 (28) | 1 (9) | 0 (0)
Weight loss (Investigations) | 1 (1) | 3 (11) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 12 (25) | 6 (19) | 2 (5) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 15 (38) | 17 (29) | 4 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (8) | 1 (1) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (8) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 10 (16) | 3 (3) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (7) | 3 (9) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (3) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (8) | 1 (3) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (4) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spasticity (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (6) | 1 (1) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (35) | 12 (24) | 4 (5) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (37) | 10 (14) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (7) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (25) | 7 (17) | 2 (2) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (6) | 4 (10) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (20) | 4 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT02443077/Prot_SAP_000.pdf
  • Informed Consent Form: PA051301_A14Consent(Untracked) (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT02443077/ICF_001.pdf
  • Informed Consent Form: PA051301_A14EarlySafetyConsent(Untracked) (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT02443077/ICF_002.pdf